CLINICAL TRIAL: NCT02170584
Title: Tolerability of Single Rising Doses of 0.1 mg, 1 mg, and 5 mg BIBR 953 ZW IV (Placebo-controlled in Each Dose Group; Substudy 1) and Absolute and Relative Bioavailability of 100mg BIBR 1048 Tablet and of Solution and of 1 mg or 5 mg BIBR 953 ZW IV (Randomized, Three-way Crossover; Substudy 2).
Brief Title: Tolerability of BIBR 953 ZW IV and Bioavailability of BIBR 1048 Tablet and Solution in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.5
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (4):
- BIBR 953 ZW IV (Experimental)
  Interventions: Drug: BIBR 953 ZW IV
- BIBR 1048 MS oral solution (Active Comparator)
  Interventions: Drug: BIBR 1048 MS oral solution
- BIBR 1048 MS tablet (Experimental)
  Interventions: Drug: BIBR 1048 MS tablet
- BIBR 953 ZW IV Placebo (Placebo Comparator)
  Interventions: Drug: BIBR 953 ZW IV Placebo

INTERVENTIONS:
Drug: BIBR 953 ZW IV
  Arms: BIBR 953 ZW IV
Drug: BIBR 1048 MS tablet
  Arms: BIBR 1048 MS tablet
Drug: BIBR 1048 MS oral solution
  Arms: BIBR 1048 MS oral solution
Drug: BIBR 953 ZW IV Placebo
  Arms: BIBR 953 ZW IV Placebo

SUMMARY:
Two substudies to assess (1) the tolerability of BIBR 953 ZW intravenous infusion at 0.1, 1 and 5 mg BIBR 953 ZW and (2) the absolute bioavailability of 100mg BIBR 1048 administered as 'acid free' tablet formulation (TF1) and (3) the bioavailability of the 100 mg tablet of BIBR 1048 relative to the tartaric acid solution of 100 mg dose strength and (4) the absolute bioavailability of the 100 mg tartaric acid solution of BIBR 1048 MS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 18 and ≤ 50 years
* Broca ≥ - 20% and ≤ + 20%

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * commotio cerebri
* Intake of drugs with a long half-life (>24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2001-01; Primary Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
AUC0-inf (Area under the plasma concentration-time curve extrapolated to infinity) | up to 48 hours after drug administration
AUC0-tf (Area under the plasma concentration-time curve up to the last quantifiable plasma concentration) | up to 48 hours after drug administration
Cmax (Maximum plasma concentration after oral administration) | up to 48 hours after drug administration
Cumulative urinary excretion of BIBR 953 ZW administered intravenously | up to 48 hours after drug administration

SECONDARY OUTCOMES:
changes in activated partial thromboplastin time (aPTT ) | up to 48 hours after drug administration
changes in prothrombin time (PT) | up to 48 hours after drug administration
C29 (Plasma concentration of BIBR 953 ZW at 29 minutes after the start of the 30 min. infusion) | 29 minutes after start of infusion
t1/2 (terminal half-life) | up to 48 hours after infusion
CLtot (total clearance of drug from plasma) | up to 48 hours after infusion
CLren (renal clearance from plasma) | up to 48 hours after infusion
MRTdisp (Mean time of residence of drug molecules in the body after intravascular administration) | up to 48 hours after infusion
Vss (apparent volume of distribution at steady state) | up to 48 hours after infusion
Vz (Apparent volume of distribution during the terminal elimination phase) | up to 48 hours after infusion
MRTtot (total mean residence time) | up to 48 hours after oral administration
CLtot/F (total clearance after oral administration) | up to 48 hours after oral administration
tmax (time to reach the peak plasma concentration) | up to 48 hours after oral administration
Vz/F (apparent volume of distribution of the terminal elimination phase after oral administration) | up to 48 hours after oral administration
changes in Ecarin clotting time (ECT) | up to 48 hours after drug administration
changes in thrombin time (TT) | up to 48 hours after drug administration
changes in vital signs (systolic and diastolic blood pressure, pulse rate) | up to 1 month
changes in electrocardiogram | up to 1 month
occurrence of adverse events | up to 1 month